CLINICAL TRIAL: NCT06406686
Title: Ablation Index in Standard vs. High Power Radiofrequency Ablation for Typical Atrial Flutter: A Randomized Study (AITAF)
Acronym: AITAF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Rory Dowd, EP fellow, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB24-0132
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Atrial Flutter; Atrial Flutter Typical; Cavotricuspid Isthmus Dependent Macroreentry Tachycardia
Keywords: Ablation; High power short duration; CARTO; QDot Micro; Ablation Index
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Single-blinded. Investigator will know study arm, patients/participants will not. The outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 Watt (Active Comparator): Power set to 30 Watts
  Interventions: Procedure: Ablation of the Cavo-tricuspid isthmus for typical Atrial Flutter
- 50 Watt (Experimental): Power set to 50 Watts
  Interventions: Procedure: Ablation of the Cavo-tricuspid isthmus for typical Atrial Flutter

INTERVENTIONS:
Procedure: Ablation of the Cavo-tricuspid isthmus for typical Atrial Flutter — Durable block across the cavotricuspid isthmus by radiofrequency ablation.

SUMMARY:
A randomized controlled trial will be conducted to evaluate the efficacy of Ablation Index-guided high power - short duration (HPSD) ablation compared to conventional power settings in Cavotricuspid Isthmus (CTI) dependent atrial flutter. Participants will be randomized to receive either AI-guided HPSD ablation at 50 Watts or conventional power settings at 30 Watts. Both arms will use the Carto 3D mapping system and the QDOT MICRO ablation catheter (Biosense Webster). An anatomically contiguous line will be created with <6mm inter-lesion distance. After a standardized wait time of 30 minutes, ablation success will be assessed. The primary outcome is total radiofrequency ablation time. Secondary outcomes include procedural time, fluoroscopy time, safety outcomes, and 3-month freedom from recurrence. It is our expectation that HPSD will result in a shorter primary outcome.

DETAILED DESCRIPTION:
Title: A Randomized Trial of Ablation Index Guided High vs Standard Power Radiofrequency Ablation for Typical Atrial Flutter

Design: Prospective, two-arm, single center, superiority study with comparison of standard 30W power settings vs 50W high power settings

Purpose: To evaluate the superiority of high-power ablation settings over standard power settings in achieving block across the CTI for typical flutter

Enrollment: A minimum of 25 subjects in each arm. Enrollment over a period of 12 months.

Subjects: Subjects referred by a cardiac electrophysiologist for standalone radiofrequency ablation of typical atrial flutter

Clinical site: Foothills Medical Center, University of Calgary, Calgary, Alberta, Canada

Endpoints: Primary endpoint: total radiofrequency time per procedure

Secondary endpoints:

RF time to initial CTI block Total procedure time Time from procedure start to procedure end Incidence of early reconnections during wait period Incidence of dormant conduction during adenosine testing Total number of ablation lesions required to achieve durable CTI block Total analgesia and sedation usage, e.g. midazolam, fentanyl and propofol in mg and/or mL Post-procedure patient perception of a) pain and b) nausea on a scale of 1 (none) to 10 (maximum possible)

Secondary safety endpoints:

Steam pops Pericardial effusions Pericardial tamponade

Secondary follow-up outcomes:

The presence of durable CTI block if a subsequent EP study is performed within 3 months of the initial procedure (e.g. AF ablation) Recurrence of documented AFL within 3 months by available ECGs, telemetry, wearable monitors, or Holters Holter at 2 months for incidence and burden of atrial arrhythmias

Materials: 3-D electro-anatomical mapping system: CARTO, Biosense Webster Diagnostic catheters: 20-pole halo catheter, 10 pole coronary sinus catheter Ablation catheter: QDOT MICRO, BiosenseWebster

Sponsors: None, fellow initiated research

Despite the existing observational data, there have been no randomized controlled trials (RCTs) investigating HPSD in CTI ablation to validate its effectiveness. Furthermore, the applicability of AI to CTI ablation has not been tested. It's important to note that CTI ablation, performed under conscious sedation, introduces respiratory movement, leading to increased CF variability, which may affect precise energy delivery.

We propose conducting the first RCT, to our knowledge, investigating the use of High-Power Short-Duration Ablation (HPSD) in the treatment of CTI-dependent flutter.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically determined by a cardiac electrophysiologist to have had at least one episode of CTI dependent atrial flutter
2. Clinically determined by a cardiac electrophysiologist likely to benefit from standalone CTI ablation
3. For this to be their first CTI ablation attempt
4. Able and willing to comply with all protocol requirements
5. Agree to and sign patient Informed Consent Form (ICF)
6. Be 18 years of age or older

Exclusion Criteria:

1. Previous CTI ablation
2. Adult congenital heart disease, including Ebstein's anomaly
3. Previous surgery involving the tricuspid valve and atrium including cannulation scars for cardiopulmonary bypass
4. Pediatric population age <18
5. Women who are pregnant or breastfeeding.
6. Active enrollment in another investigational study involving a drug or device.
7. A requirement for additional procedures in the same setting. Such as EP study and ablation of other induced arrhythmias since these prolong secondary endpoints such as procedure time and RF time
8. Patients on anti-arrhythmic drugs (AADs) such as flecainide, sotalol, or amiodarone should have their AAD stopped 3 days prior, and not be restarted after the procedure
9. Patients under General Anesthetic (GA)
10. Patients with sufficient baseline cognitive impairment to be unable to answer a post-procedure survey or consent Previous ablations, other than for CTI flutter, are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2025-06-03 (Estimated); Study Completion 2025-06-03 (Estimated)

PRIMARY OUTCOMES:
RF time to durable CTI block | End of procedure
  Cumulative delivery time of radio-frequency lesions

SECONDARY OUTCOMES:
RF time to initial CTI block | End of procedure
  At the point of initial CTI block, the total cumulative time applying radiofrequency energy
Total procedure time | End of procedure
  Time from procedure start to procedure end
Incidence of early re-connections during wait period | End of procedure
  Whether or not conduction was observed across the CTI before the wait period had expired
Total number of ablation lesions required to achieve durable CTI block | End of procedure
  At the point of durable CTI block, the total cumulative number of radiofrequency lesions deployed
Total analgesia and sedation usage | End of procedure
  Cumulative doses of sedation and analgesic medicines
Post-procedure patient perception of pain and nausea | End of procedure day
  Post-procedure patient perception of a) pain and b) nausea on a scale of 1 (none) to 10 (maximum possible) assessed after the procedure and prior to discharge.
Steam pops | End of procedure
  Count of audible "steam-pops" during the procedure
Pericardial effusions | End of procedure day
  Observation of new effusion after the procedure
Pericardial tamponade | End of procedure day
  Observation of hemodynamically significant pericardial effusion periprocedurally warranting intervention

CONTACTS AND LOCATIONS:
Overall Officials: George D Veenhuyzen, MD, Principal Investigator — University of Calgary; Rory P Dowd, MBBS, MEng, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golian M, Ramirez FD, Alqarawi W, Hansom SP, Nery PB, Redpath CJ, Nair GM, Shaw GC, Davis DR, Birnie DH, Sadek MM. High-power short-duration radiofrequency ablation of typical atrial flutter. Heart Rhythm O2. 2020 Oct 3;1(5):317-323. doi: 10.1016/j.hroo.2020.09.002. eCollection 2020 Dec. PMID 34113888